CLINICAL TRIAL: NCT06749379
Title: LIPEDEMA AWARENESS IN FIBROMYALGIA
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, MD, Ufuk University
Other Study IDs: 20/07/2022/20.478.486/1424
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia; Lipedema
Keywords: fibromyalgia, lipedema, awareness
MeSH Terms: conditions — Fibromyalgia; Lipedema | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Presence and stages of lipedema were diagnosed with examination. — Lipedema stage characteristics: stage 1: Smooth skin with a uniform increase in subcutaneous tissue; stage 2: Irregular skin surface with indentations and nodular alterations in the subcutaneous tissue; stage 3: Significant increase in circumference accompanied by loose skin/tissue ('dewlap').

SUMMARY:
Lipedema is a chronic debilitating condition that impacts the subcutaneous adipose tissue of the extremities. It is a chronic condition but should not be regarded as always progressing.The clinical course varies individually and is unpredictable. It may considerably diminish the patient's quality of life. Fibromyalgia, similar to lipedema, is a debilitating chronic pain disease of unclear origin that primarily affects women. It is a complex syndrome marked by widespread pain and tenderness. Fibromyalgia and lipedema are both marked by pain related to soft tissue. Both disorders are not amenable to curative treatment, resulting in a significant burden on individual and public health. No definitive indicators, including abnormal laboratory or imaging results, can be discerned to differentiate one disorder from another.

With this perspective, the aim of our study was to evaluate the presence of lipedema and lipedema-related factors in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* over the age of 18
* who met the fibromyalgia diagnostic criteria according to the American College of Rheumatology (ACR) 2016 Fibromyalgia Diagnostic Criteria

Exclusion Criteria:

* renal or cardiac insufficiency,
* the use of any drug that could influence body fluid and electrolyte balance,
* the presence of a major somatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study included 100 female patients over the age of 18 who met the fibromyalgia diagnostic criteria according to the American College of Rheumatology (ACR) 2016 Fibromyalgia Diagnostic Criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 1 month
  Patients were asked to mark the severity of their widespread body pain in the last week on a 10 cm visual analog scale (VAS) (0: no pain, 10: unbearable pain, the higher the measured value, the greater the pain intensity).
Presence and stages of lipedema were diagnosed according to S1 guidelines of the German Society of Phlebology | 1 month
  Overview of diagnostic criteria for lipedema; Initiation during puberty, pregnancy, or menopause, characterized by disproportionate proliferation of adipose tissue (extremities, trunk), cuffing around the joints, unaffected hands and feet, sensations of heaviness and tightness in the affected extremities, tenderness upon palpation or spontaneous pain - escalating throughout the day, edema - worsening over the course of the day, easy bruising, and a negative Stemmer's sign. Lipedema stage characteristics: stage 1: Smooth skin with a uniform increase in subcutaneous tissue; stage 2: Irregular skin surface with indentations and nodular alterations in the subcutaneous tissue; stage 3: Significant increase in circumference accompanied by loose skin/tissue ('dewlap').
The American College of Rheumatology (ACR) 2016 Fibromyalgia Diagnostic Criteria | 1 month
  It is a compilation of diagnostic criteria formulated for the identification of fibromyalgia, established following the modification of previously utilized diagnostic criteria. It comprises two components: the widespread pain index (WPI) and the symptom severity scale (SSS).
  The assessment of the WPI involves indicating persistent pain over the past seven days across five anatomical regions (upper left, upper right, lower left, lower right, axial) and 19 specific body areas (both jaws, shoulders, upper arms, lower arms, hips, upper legs, lower legs, neck, upper back, lower back, chest, and abdomen). Each region is assigned one point. The cumulative score varies from 0 to 19. For a diagnosis of widespread pain, pain must be evident in a minimum of 4 out of 5 anatomical regions.
The Revised Fibromyalgia Impact Questionnaire | 1 month
  It is a questionnaire designed to assess functional limitations and disabilities resulting from fibromyalgia. The questionnaire comprises a total of 21 questions divided into three sections: function, overall impact, and symptoms. Responses to each inquiry are indicated on a scale ranging from 0 to 10. The overall score is determined by summing the results: the score of the first section is divided by three, the score of the second section by one, and the score of the third section by two. Elevated scores signify a greater fibromyalgia-associated impairment
Beck Depression Inventory | 1 month
  It is a scale designed to assess the intensity and severity of depression symptoms. The scale comprises 21 items utilizing a 4-point Likert format, with each item rated from 0 to 3. Higher scores indicate more severe depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided